CLINICAL TRIAL: NCT04387981
Title: A Single Dose Study to Assess the Mass Balance Recovery, Absorption, Metabolism, and Excretion of [14C] Orvepitant in Healthy Male Subjects After Oral Dosing
Brief Title: Mass Balance Study of [14C]-Orvepitant Oral Solution in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nerre Therapeutics Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ORV-1-02
Record Dates: First submitted 2020-05-07; First posted 2020-05-14 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: Healthy
MeSH Terms: interventions — orvepitant

STUDY DESIGN:
Intervention Model Description: Open label, single dose
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [14C]-orvepitant (Experimental): [14C]-orvepitant administered as 30mg single dose in oral solution
  Interventions: Drug: [14C]-orvepitant

INTERVENTIONS:
Drug: [14C]-orvepitant — Oral solution of [14C]-orvepitant
  Other Names: orvepitant

SUMMARY:
This is a single centre, open-label, non-randomised study to assess the mass balance recovery, absorption, metabolism, and excretion of a single oral dose of [14C]-orvepitant in healthy male subjects. It is planned to enrol 6 subjects. Each subject will receive a single dose of 30 mg [14C] orvepitant containing not more than (NMT) 3.7 megabecquerel (MBq) [14C], administered as an oral solution in the fasted state. Subjects will be admitted in the evening on the day prior to [14C]-orvepitant administration and will be dosed in the morning following an overnight fast. It is planned that subjects will remain resident in the clinical unit until 168 hours post-dose (Day 8) when they will be discharged from the clinical unit. Through the resident period samples (blood, urine, faeces) will be collected and analysed for mass balance, total radioactivity, orvepitant levels. Metabolite profiling and ID will also be performed.

ELIGIBILITY:
Key Inclusion Criteria:

* Healthy males
* Aged 30 to 65 years inclusive at the time of signing informed consent.
* Body mass index (BMI) of 18.0 to 35.0 kg/m2 as measured at screening.
* Must provide written informed consent.
* Must agree to adhere to the contraception requirements

Key Exclusion Criteria:

* History of any drug or alcohol abuse in the past 2 years.
* Regular alcohol consumption >21 units per week.
* Current smokers and those who have smoked within the last 12 months.
* Radiation exposure, including that from the present study, excluding background radiation but including diagnostic x-rays and other medical exposures, exceeding 5 mSv in the last 12 months or 10 mSv in the last 5 years.
* Clinically significant abnormal clinical chemistry, haematology, or urinalysis as judged by the Investigator.
* Subjects with a presence of any of the following at screening: bilirubin, alanine aminotransferase (ALT), or aspartate aminotransferase (AST) >1.5 × the upper limit of normal.
* Confirmed positive drugs of abuse test result.
* Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) results.
* Evidence of renal impairment at screening, as indicated by an estimated creatinine clearance (CLcr) of <80 mL/min using the Cockcroft-Gault equation.
* History of clinically significant cardiovascular, renal, hepatic, chronic respiratory, or GI disease, neurological or psychiatric disorder, as judged by the Investigator.

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-06-28 (Actual); Study Completion 2020-06-28 (Actual)

PRIMARY OUTCOMES:
Percentage of radioactive dose recovered in urine and faeces and total percentage | 168 hours
Concentration of total radioactivity in blood and plasma | 168 hours

CONTACTS AND LOCATIONS:
Overall Officials: Principal Investigator, Principal Investigator — Quotient Sciences
Locations (1):
- Quotient Sciences, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No